CLINICAL TRIAL: NCT06452914
Title: Clinical Outcomes Related to Treatment of Distal Symmetric Polyneuropathy Using Semiconductor Embedded Therapeutic Socks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endocrine Research Solutions (Industry)
Collaborators: INCREDIWEAR HOLDINGS, INC. (Industry)
Responsible Party: Principal Investigator, John Chip H. Reed, Principal Investigator, Endocrine Research Solutions
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups; one group that will be assigned the treatment socks and the second group that will be assigned the placebo socks.
Who Masked: Participant, Investigator
Masking Description: This study is double blinded. Neither the Investigator or the subject will know which arm they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semiconductor Embedded Therapeutic Socks (Experimental): Treatment of Distal Symmetric Polyneuropathy Using Semiconductor Embedded Therapeutic Socks
  Interventions: Device: Semiconductor Embedded Therapeutic Socks
- Placebo Socks (Placebo Comparator): Treatment of Distal Symmetric Polyneuropathy Using Placebo Socks as a Comparator to Semiconductor Embedded Therapeutic Socks
  Interventions: Device: Placebo Socks

INTERVENTIONS:
Device: Semiconductor Embedded Therapeutic Socks — Semiconductor Embedded Therapeutic Socks
  Arms: Semiconductor Embedded Therapeutic Socks
Device: Placebo Socks — Socks not containing the Semiconductor Embedded Therapeutic fabric
  Arms: Placebo Socks

SUMMARY:
Distal symmetric polyneuropathy, also known as diabetic neuropathy, is the most common neurological complication of diabetes and a main cause of morbidity. The condition leads to gradual loss of function of the longest nerve fibers that limits function and decreases quality of life. Symptoms present distally and symmetrically in toes and feet. Symptoms of the neurologic disability include sensory loss, risk of foot ulcers and limb amputations and pain. The condition is not generally considered reversible, and condition management aims to slow progression and prevent complications.

According to estimates from the International Diabetes Federation, diabetic neuropathy affected approximately 425 million people in 2017, with projections indicating a rise to 628 million by 2045. Despite the high prevalence of this condition, it is commonly misdiagnosed and has limited treatment options. There are multiple phenotypes of diabetic neuropathy, with the most common form being distal symmetric sensorimotor polyneuropathy, which is what we will be focusing on in this study.

The proposed study seeks to evaluate the effectiveness of a non-compressive therapeutic socks throughout a 12-week course of rehabilitation for managing distal symmetric polyneuropathy. Outcome measures will be collected at standard intervals and compared with pre-treatment measures to evaluate effectiveness of treatment.

DETAILED DESCRIPTION:
Treatments for diabetic neuropathy includes a systematic, stepwise approach that entails glycemic control and control of metabolic syndrome, symptomatic treatment of pain, and counseling on foot care and safety measures.

Unlike compression products, the semiconductor embedded socks increase blood circulation through activation of the elements with heat of the body, and releases mid and far infrared waves as well as negative ions. Both infrared waves and negative ions are biologically active and mediate inflammatory and pain pathways in the body. The technology has also been shown to increase blood speed and blood flow. The technology has also been shown to:

* Increase blood flow and velocity
* Reduce osteoarthritis pain
* Reduce effusion post total knee arthroplasty
* Improve chondrogenic differentiation in vitro
* Improve muscle recovery
* Increase circulation by up to 22% at rest
* Improve functional outcomes

The benefits of the Infrared Wave and Negative Ion therapy include:

* Inhibition of Cox-2 and Prostaglandins in the lipopolysaccharide (LPS)-moderated pain pathway
* Up-regulation of heat shock protein
* Mediated Nitric oxide production
* Increased activity of voltage-gated ion channels
* Increased activity of mechanosensitive ion channels
* Polarization of cell surface membranes
* Protecting muscle damage
* Scavenging of Reactive Oxygen Species (ROS)
* Improved thermoregulation

To date, studies have shown that the semiconductor embedded fabric increase circulation by up to 22% at rest, and have shown powerful results in reducing inflammation, swelling, improving range of motion in the knee post-surgery, and providing pain relief.

The semiconductor embedded fabric emits mid-level and far infrared waves and negative ions. Delivery of infrared waves and negative ions to the tissue increases blood flow, facilitates the anti-inflammatory nitric oxide (NO) cascade by accelerating the binding of calcium (Ca2+) to calmodulin (CaM). NO provides several healing factors to the body as a vasodilator, increasing blood and lymphatic flow. Additionally, NO down-regulates interleukin-1 beta (IL1β) and inducible nitric oxide synthase (iNOS) in certain cell types, which leads to reduced cyclooxygenase-2 (COX-2) and prostaglandins - molecules responsible for causing inflammation and pain. Unlike other systemic COX-2 inhibitors such as nonsteroidal anti-inflammatory drugs (NSAIDs), targeted infrared and negative ion therapy stimulate localized reaction pathways, thereby reducing pain and inflammation.

This study seeks to identify patient reported outcomes for management of Diabetic Neuropathy with semiconductor embedded fabric in the affected area.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild to moderate Diabetic Neuropathy with a score between 2 and 7 out of 10 on the MNSI upon clinical examination and assessment.
* Patients reporting symptoms of Diabetic Neuropathy
* Patients age 18-79
* Patients who are willing and able to adhere to follow-up schedule and protocol guidelines
* Patients who are willing and able to sign corresponding research subject consent form

Exclusion Criteria:

* Patient has a history of neurodegenerative conditions, including multiple sclerosis or Parkinson's disease
* Patient has chronic pain conditions unrelated to diabetic neuropathy, including spinal stenosis, low back pain, and sciatica
* Patient has auto-immune or auto-inflammatory diseases other than Diabetic Neuropathy, including Multiple Sclerosis or Lyme Disease
* Patient has experienced a stroke
* Patient has any type of paralysis
* Patients with a score less than 2 and greater than 7 out of 10 on the MNSI upon clinical examination and assessment
* Patient has severe peripheral artery disease (with an ankle brachial index of <0.7)
* Patient has chronic venous insufficiency (greater than stage 4)
* Patient has used tobacco within the last 90 days
* Patient has an open wound at the area of application
* Patient has started a new medication for diabetic neuropathy symptoms within the past 90 days
* Patient is not within the ages of 18-79
* Patient is unwilling or unable to sign the corresponding research subject consent form
* Patient meets any other criteria or has any other condition that, in the opinion of the investigator, would prevent them from completing the study or that, in the opinion of the investigator, would confound study results

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Improved patient function as determined by pre-treatment and post-treatment Patient Specific Lower Extremity Functional Scale (LEFS), Michigan Neuropathy Screening Instrument (MNSI), and Quality of Life Questionnaire-Diabetic Neuropathy (QOL-DN) compared | 12 Weeks
  LEFS consists of 20 items, each scored on a 5-point scale (0 = extreme difficulty, 4 = no difficulty).
  Scoring: The maximum score is 80, with higher scores indicating better function. A lower score suggests greater disability or difficulty in performing daily activities.
  The MNSI has two parts- Part A: Self-administered questionnaire with 15 items about symptoms related to neuropathy. Scoring is based on the presence or absence of symptoms, with a higher score indicating more symptoms.
  Part B: Physical examination conducted by a healthcare professional that includes inspection of the feet and assessment of reflexes and sensation. A higher score indicates more severe neuropathy.
  QOL-DN encompasses multiple domains such as physical health, emotional well-being, social participation, and specific neurological symptoms.
  Scoring: Each domain is scored individually, and a composite score can be derived, from -4 to 136. Higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Reduction in pain as determined by pre-treatment and post-treatment Numeric Pain Rating Scale or Visual Analog Scale (VAS) compared to placebo. | 12 Weeks
  Reduction in pain as measured by Visual Analog Scale from 1 to 10, with 1 being mild and 10 being severe.
Reduction in symptom severity upon physical examination and improvement in quantitative sensory testing measures from pre-treatment measures compared to placebo. | 12 Weeks
  A series of tests are performed. Through the use of a tuning fork placed on the foot, if the patient no longer feels vibration after 8 seconds but does feel it for longer than 8 seconds when placed on the hand, severity of neuropathy can be determined. Through the use of a reflex hammer, tapping the ankle determines the presence or absence of ankle reflexes. Mono-filament testing, where after a series of touches in specific locations on the bottom of the foot, the presence or absence of sensation can be quantified.
Improvement in tissue oxygenation of the affected foot/feet as determined by clinically captured images with the non-invasive Kent Imaging device and pulse oximeter compared to placebo. | 12 Weeks
  Improvement in tissue oxygenation of the affected foot/feet as determined by clinically captured images with the non-invasive Kent Imaging device and pulse oximeter compared to placebo.
Compliance with device usage throughout the study, reported weekly. | 12 Weeks
  Device usage will be tracked with a device usage log that the patient completes based on hours the device is worn every day, to self-report compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Myers, Study Director — INCREDIWEAR HOLDINGS, INC.; John Reed, Principal Investigator — Endocrine Research Solutions. Inc.
Locations (1):
- Endocrine Research Solutions, Inc., Roswell, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is undecided if individual participant data will be made available to other researchers during or after the course of the trial.

REFERENCES:
- [Background] Roikjer J, Morch CD, Ejskjaer N. Diabetic Peripheral Neuropathy: Diagnosis and Treatment. Curr Drug Saf. 2021;16(1):2-16. doi: 10.2174/1574886315666200731173113. PMID 32735526
- [Background] Iqbal Z, Azmi S, Yadav R, Ferdousi M, Kumar M, Cuthbertson DJ, Lim J, Malik RA, Alam U. Diabetic Peripheral Neuropathy: Epidemiology, Diagnosis, and Pharmacotherapy. Clin Ther. 2018 Jun;40(6):828-849. doi: 10.1016/j.clinthera.2018.04.001. Epub 2018 Apr 30. PMID 29709457
- [Background] Csech J, Gervais C. [Aspegic]. Soins. 1982 Dec;(395-396):53-5. No abstract available. French. PMID 6820190
- [Background] Leung TK. In Vitro and In Vivo Studies of the Biological Effects of Bioceramic (a Material of Emitting High Performance Far-Infrared Ray) Irradiation. Chin J Physiol. 2015 Jun 30;58(3):147-55. doi: 10.4077/CJP.2015.BAD294. PMID 26014120
- [Background] Kyselovic J, Masarik J, Kechemir H, Koscova E, Turudic II, Hamblin MR. Physical properties and biological effects of ceramic materials emitting infrared radiation for pain, muscular activity, and musculoskeletal conditions. Photodermatol Photoimmunol Photomed. 2023 Jan;39(1):3-15. doi: 10.1111/phpp.12799. Epub 2022 May 21. PMID 35510621
- [Background] Cho SY, Roh YS, Roh HT. Evaluation of tympanic temperature and thermal sensation responses during exercise to verify the positive effects of wearing germanium-coated functional clothing. J Phys Ther Sci. 2016 Jun;28(6):1860-3. doi: 10.1589/jpts.28.1860. Epub 2016 Jun 28. PMID 27390434
- [Background] Siao P, Cros DP. Quantitative sensory testing. Phys Med Rehabil Clin N Am. 2003 May;14(2):261-86. doi: 10.1016/s1047-9651(02)00122-5. PMID 12795516
- [Background] Jia ZR, Wang TT, Wang HX. Significance of quantitative sensory testing in the diagnosis of diabetic peripheral neuropathy. J Clin Neurophysiol. 2014 Oct;31(5):437-40. doi: 10.1097/WNP.0000000000000086. PMID 25271682
- [Background] The Effect of Therapeutic Garments on Blood Flow as measured by a Laser Doppler Blood Flow Monitor; Michelle Lott, Raines DeMint. Lean RA QA Systems; May 13, 2017
- [Background] Duranti C, Bagni G, Iorio J, Colasurdo R, Devescovi V, Arcangeli A. Effects of Germanium embedded fabric on the chondrogenic differentiation of adipose derived stem cells. Tissue Cell. 2024 Oct;90:102507. doi: 10.1016/j.tice.2024.102507. Epub 2024 Jul 30. PMID 39128191
- [Background] Justice TE, Jacob PB. Non-compressive sleeves versus compression stockings after total knee arthroplasty: A prospective pilot study. J Orthop. 2023 Nov 24;49:102-106. doi: 10.1016/j.jor.2023.11.044. eCollection 2024 Mar. PMID 38094981
- [Background] Empowering Recovery: Surface Electromyography Shows how Incrediwear Helps Professional Athletes Recover. Incrediwear Holdings, Inc. Dec. 2021
- [Background] Park JH, Lee S, Cho DH, Park YM, Kang DH, Jo I. Far-infrared radiation acutely increases nitric oxide production by increasing Ca(2+) mobilization and Ca(2+)/calmodulin-dependent protein kinase II-mediated phosphorylation of endothelial nitric oxide synthase at serine 1179. Biochem Biophys Res Commun. 2013 Jul 12;436(4):601-6. doi: 10.1016/j.bbrc.2013.06.003. Epub 2013 Jun 10. PMID 23756809
- [Background] Fateh HR, Madani SP, Heshmat R, Larijani B. Correlation of Michigan neuropathy screening instrument, United Kingdom screening test and electrodiagnosis for early detection of diabetic peripheral neuropathy. J Diabetes Metab Disord. 2016 Mar 25;15:8. doi: 10.1186/s40200-016-0229-7. eCollection 2015. PMID 27019831
- [Background] NIH Repository Diabetes in Youth. Michigan Neuropathy Screening Instrument, University of Michigan 2014. https://repository.niddk.nih.gov/media/studies/search/MOPs/SEARCH%201-3%20MOP/SEARCH(16).pdf. PDF download.
- [Background] Mehta SP, Fulton A, Quach C, Thistle M, Toledo C, Evans NA. Measurement Properties of the Lower Extremity Functional Scale: A Systematic Review. J Orthop Sports Phys Ther. 2016 Mar;46(3):200-16. doi: 10.2519/jospt.2016.6165. Epub 2016 Jan 26. PMID 26813750
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Vinik EJ, Hayes RP, Oglesby A, Bastyr E, Barlow P, Ford-Molvik SL, Vinik AI. The development and validation of the Norfolk QOL-DN, a new measure of patients' perception of the effects of diabetes and diabetic neuropathy. Diabetes Technol Ther. 2005 Jun;7(3):497-508. doi: 10.1089/dia.2005.7.497. PMID 15929681
- [Background] Alghamdi M, Owolabi LF, Adamu B, Taura MG, Jibo A, Almansour M, Alaklabi SN, Alghamdi MA, Imam IA, Abdelrazak R, Rafaat A, Aliyu MH. Disease-specific quality of life in patients with diabetic neuropathy. Saudi Med J. 2022 Apr;43(4):408-417. doi: 10.15537/smj.2022.43.4.20210861. PMID 35414620
- [Background] Modi KD, Sharma AK, Mishra SK, Mithal A. Pulse oximetry for the assessment of autonomic neuropathy in diabetic patients. J Diabetes Complications. 1997 Jan-Feb;11(1):35-9. doi: 10.1016/1056-8727(95)00089-5. PMID 9025011
- [Background] Jensen MP, McFarland CA. Increasing the reliability and validity of pain intensity measurement in chronic pain patients. Pain. 1993 Nov;55(2):195-203. doi: 10.1016/0304-3959(93)90148-I. PMID 8309709
- [Background] Michael G. Sowa,